CLINICAL TRIAL: NCT02733510
Title: The Impact of Early Protocol Biopsy in Kidney Transplant Recipients Receiving TAC and MMF; a Prospective Observational Study
Brief Title: The Impact of Early Protocol Biopsy in Kidney Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Joo Kim, Professor, Samsung Medical Center
Other Study IDs: SMC 2016-02-108-002
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Renal Failure
Keywords: kidney transplantation; subclinical rejection; steroid pulse therapy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- subclinical rejection group: patients whose protocol biopsy outcome is subclinical rejection and treat with steroid pulse therapy (methylprednisolone)
  Interventions: Drug: methylprednisolone
- No rejection group: patients whose protocol biopsy outcome is normal

INTERVENTIONS:
Drug: methylprednisolone — Steroid pulse therapy : Methylprednisolone 0.5 g daily for 3 days, followed by a tapered dose of 60 mg per day for a period of five days.
  Other Names: steroid pulse therapy
  Groups: subclinical rejection group

SUMMARY:
* The purpose of this study is evaluating the impact of steroid pulse therapy (SPT) on SCR revealed on PB in KT recipients maintained on TAC/MMF and corticosteroid.
* In our institution, since routine protocol biopsies are performed at 2 weeks, 1 year, and 2 years after renal transplantation, it is practically difficult that graft survival is used as an endpoint for randomized controlled trials.
* From a meta-analysis for 31 observational studies , acute rejection was associated with an increased risk of graft loss risk ratios ranged from 1.2 - 10.5. Furthermore, chronic allograft nephropathy and graft survival is strongly correlated with acute rejection episode during the first year after renal transplantation.
* Therefore, the aim of this study is to investigate the effect of early steroid pulse therapy for the reduction of acute rejection episode during the first year after KT in the patients who will show subclinical changes at 2-week protocol biopsy.
* The histological feature at 1 year PB, graft function (represented by serum creatinine level and eGFR) during the 1st year of KT were compared between SCR group and non-SCR group.
* Additional benefits including early detection of polioma BK virus associated nephritis (BKVAN) and relapsed underlying disease are also evaluated.

DETAILED DESCRIPTION:
* All recipients will receive induction therapy with basiliximab or rATG and triple maintenance immunosuppression with TAC/MMF and corticosteroid.
* PB at 2 weeks and 1 year after transplantation will be performed using an 18-gauge needle under ultrasound guidance.
* Patients who will get PB can be the candidate of this study.
* Methylprednisolone 0.5 g daily for 3 days will be administered in patients with SCR.
* Information of enrolled patient including age, sex, height, body weight, serum creatinine level, modality of dialysis, duration of dialysis, panel reactive antibody, donor specific antibody, HLA mismatch, ABO incompatibility and history of previous transplantation will be collected. These data will be safely controlled by the person in charge. Patient name will be changed in to initials and registration number of hospital will be changed into new registration number of this study.
* laboratory tests including WBC, BUN, creatinine, FK level, MPA level, CMV virus DNA load, BK virus DNA load, urine nitrate, urine leukocyte esterase, urine BK virus DNA load, urine culture and chest X-ray will be checked on 14th post-operative day and every month until 1year after KT.
* Enrolled patients will be followed for 1 year and routinely undergo 1-year protocol biopsy.
* Within 1 year follow up period, clinical biopsy is performed when recipients' serum creatinine level raised more than 25% of baseline level.
* The primary end point
* Biopsy proven acute rejection event within 1 year after renal transplantation
* Histologic feature including persistent SCR (the presence of SCR at both 2-week and 1-year protocol biopsy), chronic nephropathy at 1-year protocol biopsy.
* Graft kidney function estimated by serum creatinine level and eGFR
* The incidence of opportunistic infection including pneumonia, urinary tract infection, tuberculosis, fungal infection, and viral infections (such as cytomegalo, polyoma, and parvo-virus) within 1 year
* Secondary end points include effect of early detection of polioma BK virus associated nephritis (BKVAN) and relapsed underlying disease

ELIGIBILITY:
Inclusion Criteria:

* Age 19 - 70 years.
* The patients who underwent renal transplantation.
* The patients who will show rejection in 2-week protocol biopsy with stable graft function will be included in this study.

  * Stable function is defined as serum creatinine ≤1.5 mg/dl and ≤15% increase in serum creatinine in the 2 weeks before biopsy.

Exclusion Criteria:

* The patients who had clinical uremic symptom within 2 weeks after kidney transplantation..
* The patients who had elevated serum creatinine level more than 1.5mg/dl or 15% compared to previous result.
* The patients' age under 19 years or over 70 years.
* The patients who underwent preoperative desensitization.
* The patients who had multiple organ transplantation.
* The patients who showed an allergic reaction to steroid.
* The patients who had psychologic disease (eg. depression) or history of psychologic medication.
* The patients who did not agree with a consent form.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: kidney transplantation recipients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
biopsy proven acute rejection event | within 1 year after renal transplantation
incidence of opportunistic infection | within 1 year after renal transplantation

SECONDARY OUTCOMES:
histologic feature at 1 year protocol biopsy | 1 year after renal transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sung Joo Kim, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Organ Transplant Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Rush D, Nickerson P, Gough J, McKenna R, Grimm P, Cheang M, Trpkov K, Solez K, Jeffery J. Beneficial effects of treatment of early subclinical rejection: a randomized study. J Am Soc Nephrol. 1998 Nov;9(11):2129-34. doi: 10.1681/ASN.V9112129. PMID 9808101
- [Result] Gloor JM, Cohen AJ, Lager DJ, Grande JP, Fidler ME, Velosa JA, Larson TS, Schwab TR, Griffin MD, Prieto M, Nyberg SL, Sterioff S, Kremers WK, Stegall MD. Subclinical rejection in tacrolimus-treated renal transplant recipients. Transplantation. 2002 Jun 27;73(12):1965-8. doi: 10.1097/00007890-200206270-00023. PMID 12131699
- [Result] Shishido S, Asanuma H, Nakai H, Mori Y, Satoh H, Kamimaki I, Hataya H, Ikeda M, Honda M, Hasegawa A. The impact of repeated subclinical acute rejection on the progression of chronic allograft nephropathy. J Am Soc Nephrol. 2003 Apr;14(4):1046-52. doi: 10.1097/01.asn.0000056189.02819.32. PMID 12660340
- [Result] Choi BS, Shin MJ, Shin SJ, Kim YS, Choi YJ, Kim YS, Moon IS, Kim SY, Koh YB, Bang BK, Yang CW. Clinical significance of an early protocol biopsy in living-donor renal transplantation: ten-year experience at a single center. Am J Transplant. 2005 Jun;5(6):1354-60. doi: 10.1111/j.1600-6143.2005.00830.x. PMID 15888041
- [Result] Miyagi M, Ishikawa Y, Mizuiri S, Aikawa A, Ohara T, Hasegawa A. Significance of subclinical rejection in early renal allograft biopsies for chronic allograft dysfunction. Clin Transplant. 2005 Aug;19(4):456-65. doi: 10.1111/j.1399-0012.2005.00303.x. PMID 16008588
- [Result] Cosio FG, El Ters M, Cornell LD, Schinstock CA, Stegall MD. Changing Kidney Allograft Histology Early Posttransplant: Prognostic Implications of 1-Year Protocol Biopsies. Am J Transplant. 2016 Jan;16(1):194-203. doi: 10.1111/ajt.13423. Epub 2015 Aug 14. PMID 26274817
- [Result] Nickerson PW, Rush DN. Begin at the Beginning to Prevent the End. J Am Soc Nephrol. 2015 Jul;26(7):1483-5. doi: 10.1681/ASN.2014111115. Epub 2015 Jan 2. No abstract available. PMID 25556171
- [Result] Loupy A, Vernerey D, Tinel C, Aubert O, Duong van Huyen JP, Rabant M, Verine J, Nochy D, Empana JP, Martinez F, Glotz D, Jouven X, Legendre C, Lefaucheur C. Subclinical Rejection Phenotypes at 1 Year Post-Transplant and Outcome of Kidney Allografts. J Am Soc Nephrol. 2015 Jul;26(7):1721-31. doi: 10.1681/ASN.2014040399. Epub 2015 Jan 2. PMID 25556173